CLINICAL TRIAL: NCT02645201
Title: Effect of a Probiotic Combination (Gastrus®) on Adverse Effects of Therapy and on Eradication Rate of Helicobacter Pylori Infection in Children
Brief Title: The Effect of Probiotic Combination on Helicobacter Pylori Infection in Children
Acronym: Gastrus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The research protocol was completely changed.
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tadej Battelino, Prof.dr. Tadej Battelino, MD PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gastrus01
Record Dates: First submitted 2015-12-12; First posted 2016-01-01 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Helicobacter Infections
Keywords: probiotic
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Children in probiotic group will receive chewable tablets containing 4x108 CFU of Gastrus. Subjects will take 1 tablet twice a day for 21 days
  Interventions: Dietary Supplement: Gastrus
- Placebo (Placebo Comparator): Children in placebo group will receive placebo tablets of similar appearance and taste as Gastrus tablets. Subjects will take 1 placebo tablet twice a day for 21 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gastrus — to compare Gastrus 4x108 tbl twice a day to placebo tbl
  Other Names: Lactobacillus reuteri (ATC 55730 and ATCC PTA 6457)
  Arms: Probiotic
Other: Placebo — to compare Gastrus 4x108 tbl twice a day to placebo tbl
  Other Names: Placebo pills
  Arms: Placebo

SUMMARY:
The combination of two Lactubacillus reuteri strains, ATC 55730 and ATCC PTA 6457 are marketed as GASTRUS® and has been proposed as better option in increasing Helicobacter pylori eradication rate compared to the single strain ATC 55730, due to additional anti-inflammatory properties of the second strain.

Objectives of the study are to determine whether adding probiotic combination (GASTRUS®) to an anti- Helicobacter pylori regimen decreases adverse events and increases the eradication rate of Helicobacter pylori in the pediatric population infected with Helicobacter pylori bacteria.

DETAILED DESCRIPTION:
This is a 10 week, randomized, double blind, placebo controlled, multicenter study to evaluate the efficacy of GASTRUS® on the frequency of adverse events and eradication rate of H. pylori infection in children.

Subjects: Children aged 5 (>15 kg) -18 years, diagnosed with H. pylori infection during upper endoscopy with at least two validated tests, who meet all inclusion and exclusion criteria listed below. Subjects who are RUT (Rapid Urease Test) positive on the day of endoscopy will be offered to participate in the study, which includes 3 visits. They will be given information about the study and a 1-week diary to be filled out before visit 1. The properly filled diary will be considered as the screening tool to include the patients into the study and will be also considered as part of the study. At visit 1 written informed consent must be obtained from the caregivers and also from participants above 10 years of age. At each visit, physical examination will be performed as well as symptom assessment and diary evaluation. Only patients who have a positive culture for H. pylori and antibiotic susceptibility testing with no double resistance, and have filled in the diary will be enrolled. Patients will receive a prescription for triple therapy: omeprazole, amoxicillin and metronidazole / clarithromycin for 14 days depending on the antibiotic susceptibility. The dose regimens will be determined according to the weight of the child. The children will be randomized to receive chewable tablets containing 4x108 CFU of GASTRUS® or placebo of similar appearance and taste. Active and placebo tablets will be supplied. Subjects will take 1 tablet twice a day for 21 days. Diary 2 - will be dispensed (with instructions) and filled for 21 days until visit 2. Visit 2 will take place 21+/- 3 days after visit 1. At this visit a physical exam will be performed and diary 2 will be collected. Diary 3 will be reminded to be filled out one week before visit 3 which will be planned 8 weeks after visit 2 +/- 5 days. At visit 3, diary 3 will be collected. 13C-urea breath test or monoclonal stool antigen test will be performed to assess the H. pylori status after eradication treatment. In order to ensure that the children will fill their diaries, the parents will be phoned one week before visit 2 and 3.

Our study population will be children from all over Europe and Israel diagnosed with H. pylori infection with at least two recommended diagnostic methods. The investigators will complete documents considered for enrolment.

The sample size was calculated assuming that adverse effects will develop in 30% of treated children, aiming to detect difference of 20% based on a 0.80 power to detect statistically significant difference; therefore the recruitment will continue until 118 subjects are randomized into the 2 groups (test and placebo) of at least 59 children each. The estimated time to finish the study is 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Either sex age between 5 (>15 kg) - 18 years.
2. Confirmed H. pylori infection (two out of four invasive methods positive (rapid urease test/histology/culture/PCR test) with positive culture and susceptibility testing for clarithromycin and metronidazole).
3. Able to be informed (patient/parents) of the nature of the study and willing to give written informed consent (consent from the parents must be obtained before any study-related procedures are conducted and assent of the child if older than 10 years).
4. Treatment naive children with H. pylori infection.

Exclusion Criteria:

1. Significant acute or chronic GE disease (IBD, symptomatic coeliac disease…)
2. Known allergies to used antibiotics, proton pump inhibitors or probiotics
3. Having received treatment with antibiotics or bismuth compounds during the previous 30 days before endoscopy.
4. Having received proton pump inhibitors during the previous two weeks.
5. Having received probiotic therapy during the previous 14 days.
6. Being infected with a strain resistant to clarithromycin and metronidazole (double resistant)
7. Severe acquired or primary immunodeficiency.
8. Children with gastric or duodenal peptic ulcer disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-18 (Estimated); Study Completion 2017-08-18 (Estimated)

PRIMARY OUTCOMES:
to compare changes of frequency and type of adverse events (abdominal pain, duration of pain, nausea, heartburn, vomiting, taste disturbance, stool consistency) in probiotic and placebo arm at different time frames | at visit 1, visit 2 (after 3 weeks), visit 3 (after 8 weeks)
  symptom diary (abdominal pain, duration of pain, nausea, heartburn, vomiting, taste disturbance, stool consistency-frequency)

SECONDARY OUTCOMES:
to compare the number of patients with succesful eradication of Helicobacter pylori infection in probiotic and placebo arm | 8-12 weeks after eradication therapy
  13C-urea breath test or monoclonal stool antigen test

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Homan, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (5):
- Queen Fabiola Children's Hospital, Brussels, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- Dr. von Hauner Children's Hospital, Munich, Germany
- Kaplan Medical Center, Rehovot, Israel
- University Children's Hospital, Ljubljana, Slovenia

REFERENCES:
- [Result] Francavilla R, Polimeno L, Demichina A, Maurogiovanni G, Principi B, Scaccianoce G, Ierardi E, Russo F, Riezzo G, Di Leo A, Cavallo L, Francavilla A, Versalovic J. Lactobacillus reuteri strain combination in Helicobacter pylori infection: a randomized, double-blind, placebo-controlled study. J Clin Gastroenterol. 2014 May-Jun;48(5):407-13. doi: 10.1097/MCG.0000000000000007. PMID 24296423